CLINICAL TRIAL: NCT05616117
Title: Next-generation Effects of Vitamin D Supplementation in Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 01092022
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-10

CONDITIONS: Growth; Vitamin D Supplementation; Immune System Diseases; Child Development
MeSH Terms: conditions — Immune System Diseases | interventions — Cholecalciferol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We are collecting bloodsamples at birth and after one year. Further we collect meconium-samples at birth
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High-dose intrauterine D3-vitamin: Children of mothers who received 90 µg vitamin D3 daily during pregnancy from 12 weeks to delivery.
  Interventions: Other: Intrauterine 90µg D-vitamin
- Low-dose intrauterine D3-vitamin: Children of mothers who received 10 µg vitamin D3 daily during pregnancy from 12 weeks to delivery
  Interventions: Other: Intrauterine 10µg D-vitamin

INTERVENTIONS:
Other: Intrauterine 90µg D-vitamin — Children of mothers who received 90 µg vitamin D3 daily during pregnancy:10 µg from a standard prenatal multivitamin + an additional supplement containing 80µg of vitamin D3
  Groups: High-dose intrauterine D3-vitamin
Other: Intrauterine 10µg D-vitamin — Children of mothers who received 10 µg vitamin D3 daily during pregnancy, which is the dose in a standard prenatal multivitamin and the dose currently recommended by the Danish Health Authorities to all pregnant women. They will receive a prenatal vitamin containing 10µg of vitamin D + a placebo supplement.
  Groups: Low-dose intrauterine D3-vitamin

SUMMARY:
Vitamin D deficiency is common among pregnant women, despite daily vitamin D supplements. This study aims to investigate if maternal vitamin D intake of 90 vs 10 µg affects the overall health, growth, and immune system of the offspring at birth and after 1 year. Blood samples at birth and after one year, questionnaires and clinical 1-year examination will be performed on the children.

DETAILED DESCRIPTION:
Vitamin D deficiency is common among Danish pregnant women, although most pregnant women adhere to guidelines of a daily supplement of 10 µg vitamin D. Vitamin D deficiency increases the risk of complications in the pregnancy e.g., preeclampsia, gestational diabetes mellitus and fetal growth retardation. Several studies indicate that the offspring has an increased risk of immune diseases e.g., asthma and autoimmune related diseases e.g., multiple sclerosis if the mother had vitamin D deficiency during the pregnancy. It is well known that vitamin D affects the immune system, which raises the question of the effects of vitamin D supplements and which doses to give optimally.

This study aims to investigate if maternal vitamin D intake of 90 vs 10 µg D3 affects the overall health, growth, and immune system of the offspring at birth and after 1 year. Blood samples at birth and after 1 year, questionnaires and clinical 1-year examination will be performed on the children. The hypothesis is that increased vitamin D supplementation in pregnancy improves fetal development including the offspring's immune system and the developing brain. The effects of vitamin D supplementation will strengthen the offspring's overall health at birth and during their first year of life. Hopefully, this can, in the future, be part of a guideline to which dose of vitamin D is recommended for Danish pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Born by mother from our previous RCT (NCT04291313)
* All with parental authority have given consent for inclusion

Exclusion Criteria:

* Mother with compliance <80% to study drug
* Mother has denied further contact in this follow-up study

Max Age: 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children born to mothers participated in our previous RCT (NCT04291313)
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Growth of child | From birth to 11-13 month of age
  The growth from birth to the clinical examination at 11-13 month of age
Immune cell function | From birth to 11-13 month of age
  The immune cell function at birth and at 11-13 month of age.

SECONDARY OUTCOMES:
Well-being and developmental scores | At birth and at 11-13 month of age
  ASQ-3 scores and parent-reported well-being of the children at 11-13 month of age.
Hospital contact | At birth to 11-13 month of age
  Number of hospital contacts during the first year
Parent reported infections | At birth to 11-13 month of age
  Number of infections during the first year of life
Colic | At birth to 11-13 month of age
  Does the child have colic
Medicine use | At birth to 11-13 month of age
  Parent reported use of medicine, incl. astma-medicine and movicol.
Scanning of the anterior fontanelle | At 11-13 month of age.
  Ultrasound-scan of the anterior fontanelle

CONTACTS AND LOCATIONS:
Overall Officials: Pinar Bor, MD, PhD, Principal Investigator — Department of Obstetrics and Gynaecology, Regional Hospital Randers

IPD SHARING:
Plan to Share IPD: No